CLINICAL TRIAL: NCT02222792
Title: Evaluation of the BJI Inoplex 2 Kit for the Multiplex Serological Diagnosis of Bone and Joint Prosthetic Device Infections
Brief Title: BJI Inoplex 2 : Test for Diagnosis of Prosthetic Infections
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Diaxonhit (Industry)
Responsible Party: Sponsor
Other Study IDs: BJI 2
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Bone and Joint Prosthetic Infections
Keywords: Staphylococci, Streptococci, P acnes and Gram-negative bacteria

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serologic assays of sera collected from septic or non-septic patients will be performed in series and operators will be blind in terms of clinical and microbiological status in order to avoid any interpretation bias due to information collected in advance
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Septic patient group: The septic patient group will be comprised of patients presenting with bone and joint prosthetic device infection confirmed by intraoperative microbiological culture (at least 2 deep positive samples for the same bacterial strain).
- Non-septic patient group: The non-septic patient group will be comprised of prosthetic patients presenting with symptoms of mechanical loosening, and whose deep intraoperative samples have all proved negative
- Intermediate group: An intermediate group will be comprised of patients with only one deep positive sample.

SUMMARY:
A national, prospective, open-label, non-interventional, multicentre, controlled study designed to evaluate a diagnostic method in patients undergoing hip, knee or shoulder prosthetic removal regardless of whether or not infection is suspected. Serological test results will have no impact on the therapeutic approach.

Study objective: To evaluate the diagnostic performance of an antibody detection kit for the serological diagnosis of bone and joint prosthetic device infections cause by Staphylococci, Streptococci, Propionibacterium acnes (P. acnes) and Gram-negative bacteria versus the reference method: the bacterial culture of deep intraoperative samples.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. Patients 18 years of age or older
3. Patient with a bone and joint prosthetic device: total hip prosthesis (THP) or total knee prosthesis (TKP) or total shoulder prosthesis (TSP)
4. Patients with a revision of a failed prosthesis, regardless of the cause and whether septic or not
5. Patients who have not expressed their opposition to the use of their personal medical data and blood samples

Exclusion Criteria:

1. Patients already enrolled or clinically reviewed following a relapse
2. Patients with several prostheses requiring at least two revisions during the same surgical procedure
3. Patients for whom the microbiologist and/or doctor responsible for the care refuses that these patients participate in the study
4. HIV+ patients
5. Patients undergoing chemotherapy for a blood disease or solid tumour
6. Patients under guardianship or trusteeship
7. Patients who are expected to be difficult to monitor (life expectancy less than 1 year, or homeless people, foreigner in transit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The septic patient group will be comprised of patients presenting with bone and joint prosthetic device infection confirmed by intraoperative microbiological culture (at least 2 deep positive samples for the same bacterial strain).
  The non-septic patient group will be comprised of prosthetic patients presenting with symptoms of mechanical loosening, and whose deep intraoperative samples have all proved negative.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of test BJI 2 | 2 years
  The diagnostic performance of the test during unique titration.
  * Sensitivity: estimated from the proportion of septic group patients with an antibody level above the defined threshold antibody concentration.
  * Specificity: estimated from the proportion of non-septic-group patients with an antibody level less than or equal to the defined threshold antibody concentration.
  * Positive likelihood ratio.
  * Negative likelihood ratio.

SECONDARY OUTCOMES:
Interest of test BJI 2 | 2 years
  * To evaluate the diagnostic interest of the BJI Inoplex 2 test in conjunction with the clinical and laboratory data collected: diagnostic strategy and score combining several criteria.
  * To evaluate the potential medical and economic benefits of using the test: number and cost of joint aspirations or hospital stays that would have been avoided, delayed diagnosis.
  * To describe the serological outcome after surgery in septic patients.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Groupe hospitalier Diaconesses Croix Saint Simon, Paris